CLINICAL TRIAL: NCT06262139
Title: An Open-label Evaluation of a Targeted Magnetic Resonance Imaging Contrast Agent (MT218) in Prostate Cancer Patients
Brief Title: Evaluation of a Targeted Magnetic Resonance Imaging Contrast Agent in Prostate Cancer Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Songqi Gao (Industry)
Collaborators: Emory University (Other)
Responsible Party: Sponsor-Investigator, Songqi Gao, Principal investigator and Vice president, Molecular Theranostics LLC
Organization: Molecular Theranostics LLC (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: MT218-002
Record Dates: First submitted 2024-01-23; First posted 2024-02-15 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: MRI Scan
Keywords: MT218; target GBCA; peptide; MRI contrast agent; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: prostate cancer patients
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MT218 (Experimental): Each patient will receive a single intravenous injection of MT218 while being scanned with standard MR imaging sequences/protocol. The first cohort of four subjects will receive 0.02 mmol/kg, second cohort of four subjects will receive 0.04 mmol/kg, and third cohort of four subjects will receive 0.06 mmol/kg of MT218.
  Interventions: Drug: MT218 injection

INTERVENTIONS:
Drug: MT218 injection — a targeted magnetic resonance imaging contrast agent

SUMMARY:
This phase 1b open label, dose-escalating investigation study is to evaluate the dose dependent initial efficacy of the use of MT218 injection for biomarker targeted MR molecular imaging (MRMI) of prostate cancer in patients scheduled for radical prostatectomy.

DETAILED DESCRIPTION:
Phase 1b open label, single-arm, dose-escalating investigation of safety and efficacy of a gadolinium (Gd) and peptide based MRI contrast agent (MT218) as an extradomain-B fibronectin (EDB-FN) targeted molecular MR contrast agent to detect aggressive prostate cancer with comparison of its results with the standard-of-care mutliparametic MRI (mpMRI) and PSMA PET/CT and histopathology validation in preprostatectomy patients diagnosed with prostate cancer in their clinical care.

ELIGIBILITY:
Inclusion criteria

* Male subjects aged >18 years.
* Patients with confirmed Gleason score of 8 - 10 prostate cancer, had at least one prostate mpMRI and one prostate biopsy.
* Ability to lie still for MRI scanning.
* Patients must be able to provide written informed consent.
* Glomerular filtration rate (GFR) > 60 mL/min within a 30 days of the research MRI.

Key exclusion criteria

* Any diagnosis of active acute, chronic, or sub-chronic kidney or liver disease.
* Documented acute prostatitis, symptomatic or severe benign prostatic hyperplasia (BPH) or urinary tract infections.
* Patients with uncontrolled diabetes or hypertension.
* Patients with active non-prostate malignancy.
* Patients with contraindications for MRI including implantable pace makers, cochlear implants.
* Patients with uni- or bilateral hip prosthesis.
* Subjects with other significant medical conditions that would create unacceptable operative risk, compromise retention on study or compromise study related assessments.
* Major surgery within 4 weeks prior to entry on this study or patients who have not recovered from side effects of such therapy.
* Prostate biopsy within 4 weeks prior to entry on this study in which inflammation might affect MRI result.
* Subjects who received or will receive any other MRI contrast agent within 48 hours prior to MT218 injection or up to 24 hours after MT218 injection.
* Is determined by the investigator that the patient is clinically unsuitable for the study.
* Is incapable of understanding the language in which the information for the patient is given.
* Participation in a concurrent clinical trial or in another trial within the past 30 days.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Detection of aggressive prostate cancer (Gleason score 8 to 10) using peptide based MRI contrast agent (MT218) with comparing the previous clinical mpMRI using the clinical standard MRI contrast agent and PSMA-PET/CT | up to 3 days after injection
  Gleason scoring is the most common prostate cancer grading system. A Gleason score of 6 is a low-grade cancer. A Gleason score of 7 is a medium-grade cancer, and a score of 8, 9 or 10 is a high-grade cancer.
  mpMRI: multi-parametric MRI; PSMA-PET/CT: prostate-specific membrane antigen (PSMA) Positron Emission Tomography (PET) and Computed Tomography (CT) scan

CONTACTS AND LOCATIONS:
Overall Officials: David Schuster, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Evaluation of Physicochemical Properties, Pharmacokinetics, Biodistribution, Toxicity, and Contrast-Enhanced Cancer MRI of a Cancer-Targeting Contrast Agent, MT218 — http://pubmed.ncbi.nlm.nih.gov/35703463/